CLINICAL TRIAL: NCT04099940
Title: Virtual Reality Avatar Therapy for People Hearing Voices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Stephan T. Egger, Senior Psychiatrists, Psychiatric University Hospital, Zurich
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: VRAT- ATP
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Psychosis; Schizophrenia; Schizo Affective Disorder; Hearing Voices When No One is Talking (Symptom)
Keywords: Hearing Voices, Virtual Reality Avatar Therapy, Cognitive Behavioural Therapy
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Hallucinations

STUDY DESIGN:
Intervention Model Description: The investigators plan to conduct a single-blind, randomised, controlled trial in a cross-over design to assess the feasibility and efficacy of VRAT in patients with acoustic hallucinations, independent of the main diagnosis.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Avatar Therapy (VRAT) (Experimental): In the VRAT, patients with schizophrenia and acoustic hallucinations design a visual and auditory recreation (avatar) of the entity to which they attribute their hallucinations. Working with a therapist over the course of several sessions, participants change the avatar from controlling to benevolent.
  Interventions: Behavioral: Virtual Reality Avatar Therapy (VRAT); Behavioral: Assertiveness Training Program (ATP)
- Assertiveness Training Program (ATP) (Active Comparator): The ATP is a transdiagnostic cognitive behavioural treatment programme, which aims to increase self-confidence and social competence in patients with a psychiatric disorder.
  Interventions: Behavioral: Virtual Reality Avatar Therapy (VRAT); Behavioral: Assertiveness Training Program (ATP)

INTERVENTIONS:
Behavioral: Virtual Reality Avatar Therapy (VRAT) — The Virtual Reality Avatar Therapy (VRAT) is a Cognitive Behavioral Intervention, delivered through Virtual Reality.
Behavioral: Assertiveness Training Program (ATP) — The Assertiveness Training Program (ATP) is a Cognitive Behavioral Intervention, delivered as group therapy.

SUMMARY:
Hearing voices is probably the worst form of acoustic hallucinations; which can be experienced as severely disturbing and is influenced by diverse factors including the ability of the individual to influence and control the hallucinatory experience itself. In recent years virtual reality has become a treatment option. In the so-called AVATAR Therapy, patients with schizophrenia and acoustic hallucinations design a visual and auditory recreation (avatar) of the entity to which they attribute their hallucinations. Working with a therapist over the course of several sessions, participants change the avatar from controlling to benevolent. Avatar Therapy involves similar processes to learning and cognitive restructuring, comparable to other psychotherapeutic interventions. The investigators plan to conduct an interventional study using a cross-over design, to compare the feasibility and efficacy of virtual reality avatar therapy for patients with acoustic hallucinations (independent of psychiatric diagnosis) with a cognitive behavioural group therapy aimed to improve social competence.

ELIGIBILITY:
Inclusion Criteria:

* Consistent acoustic hallucinations, with the presence of voices for at least two months.
* Participants are competent to give informed consent, as determined by the referring physician or psychiatrist.
* German language proficiency as a native speaker or level B1 Common European Framework of Reference for Languages (CEFRL)

Exclusion Criteria:

* Current neurological disorder.
* Current substance use or withdrawal.
* Concomitant group psychotherapeutic intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychopathological Assessment | Change: Baseline, 3, 6 weeks, 6 and 12 months]
  Symptom Questionnaire

SECONDARY OUTCOMES:
Psychotic Symptoms | Change: Baseline, 3, 6 weeks, 6 and 12 months]
  Symptom Questionnaire
Insecurity- Self-confidence | Change: Baseline, 3, 6 weeks, 6 and 12 months]
  Symptom Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatrische Universitätsklinik Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craig TK, Rus-Calafell M, Ward T, Leff JP, Huckvale M, Howarth E, Emsley R, Garety PA. AVATAR therapy for auditory verbal hallucinations in people with psychosis: a single-blind, randomised controlled trial. Lancet Psychiatry. 2018 Jan;5(1):31-40. doi: 10.1016/S2215-0366(17)30427-3. Epub 2017 Nov 23. PMID 29175276
- [Derived] Brander M, Egger ST, Hurlimann N, Seifritz E, Sumner RW, Vetter S, Magnenat S. Virtual Reality Human-Human Interface to Deliver Psychotherapy to People Experiencing Auditory Verbal Hallucinations: Development and Usability Study. JMIR Serious Games. 2021 Jun 1;9(2):e26820. doi: 10.2196/26820. PMID 33769295